CLINICAL TRIAL: NCT03281694
Title: The Use of AVL-3288 to Potentiate the Attention-Enhancing Effects of Low-Dose Nicotine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supplier did not come through.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Professor, Director Maryland Psychiatric Research Center, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-0009999
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Change
Keywords: nicotine; positive allosteric modulator; attention; cognition
MeSH Terms: interventions — Nicotine; AVL3288

STUDY DESIGN:
Masking Description: The study will be double-blind. Only the statistician performing randomization and the dispensing pharmacist will know the sequence of test conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine - AVL-3288 Interaction Study (Other): Over four different test days, all participants will be tested with Placebo, Nicotine, AVL-3288, and Nicotine + AVL-3288, in a counterbalanced sequence.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: AVL-3288; Drug: Nicotine + AVL-3288

INTERVENTIONS:
Drug: Placebo — placebo skin patch and placebo oral solution
Drug: Nicotine — nicotine skin patch (7 mg/24 hrs) and placebo oral solution
Drug: AVL-3288 — placebo skin patch and AVL-3288 oral solution (3 mg)
Drug: Nicotine + AVL-3288 — nicotine skin patch (7 mg/24 hrs) and AVL-3288 oral solution (3 mg)

SUMMARY:
Single-center, randomized, double-blind, placebo-controlled, proof-of-principle study to evaluate potential cognitive benefits of a single oral dose of AVL-3288 (3 mg) in the presence and absence of transdermal nicotine (7 mg/24 hrs) in healthy non-smokers, while monitoring the safety and tolerability of AVL-3288.

DETAILED DESCRIPTION:
Nicotinic acetylcholine receptor (nAChR) agonists such as nicotine have been shown to enhance cognitive performance, especially functions in the attention domain. Efforts have been made to develop similar compounds as therapeutic agents for disorders such as schizophrenia or Alzheimer's disease. Over the last two decades, drug development has invested into novel nAChR agonists. Effects have generally been in the expected direction, but tended to be of small magnitude. A potential way of increasing the effect size ceiling is by co-administering a nAChR positive allosteric modulator (PAM). PAMs generally do not activate the nAChR on their own but bind to a second, modulatory site and facilitate agonist-induced responses. The present study is aimed at testing the effects of AVL-3288, a PAM selective for the α7 nAChR subtype that is thought to be of particular relevance for cognition in schizophrenia, on cognitive task performance, and on nicotine-induced improvements in cognitive task performance, in healthy adult non-smokers.

The aim of the present study is to provide the proof-of-principle that the attention-enhancing effects of the prototypical nAChR agonist nicotine can be potentiated by an α7 nAChR PAM (AVL-3288). Potentiation of nAChR agonist effects by PAMs have been shown in preclinical behavioral assays. The availability of AVL-3288 as a safe pure nAChR PAM for human research allows testing the hypothesis that nicotine and AVL-3288 will have additive or synergistic effects, such that the attention-enhancing effects of nicotine and AVL-3288 combined will be greater than the effects of either drug alone.

AVL-3288 has shown preclinical efficacy in rat paradigms of attention and memory, including models of cognitive dysfunction1-3. A human study in healthy adults reported no adverse effects associated with AVL-3288, tested at doses of 3, 10, and 30 mg. Some of the participants tested with 3 mg were smokers, some on nicotine replacement.

The present study will adopt a repeated measures design, in which a single group of 24 healthy non-smokers will complete 4 test sessions, in each of which they perform the same three cognitive paradigms. In each session, a skin patch will be administered 5 hrs prior to testing, and a solution (3 mL) will be administered by mouth 1 hr prior to testing. The skin patch is either a 7 mg/24 hrs nicotine patch or a placebo patch. The solution either contains AVL-3288 (3 mg) or is inactive diluent only. Over the 4 test sessions, each participant will be tested with Placebo + Placebo, Nicotine + Placebo, Placebo + AVL-3288, and Nicotine + AVL-3288, in a 2x2 factorial design. The sequence of test conditions will be only known to the statistician and pharmacist and counterbalanced across subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-50 years.
* Male or female willing to use qualified methods of contraception for the study duration and up to 2 months after its end. Qualified methods are: intrauterine device, condoms, oral contraceptives, surgical sterilization of the subject or the partner at least one year in advance, or postmenopausal status of the female defined as at least two years without menstruation.
* No exposure to any nicotine-containing product in the last year.
* Smoked no more that 40 cigarettes, cigars or cigarillos in lifetime.
* Normal or corrected to normal vision (at least 20/80).
* Body weight 110-220 lbs.

Exclusion Criteria:

* Pregnant or breast-feeding.
* DSM Axis I mood, anxiety or psychotic disorder.
* Drug or alcohol abuse or dependence currently or in the last 2 years.
* Cardiovascular or cerebrovascular disease, such as history of myocardial infarction and ischemia, heart failure, angina, stroke, severe arrhythmias, or EKG abnormalities (see below).
* Uncontrolled hypertension (resting systolic BP >150 or diastolic >95 mm Hg).
* Hypotension (resting systolic BP below 90 or diastolic below 60).
* Significant kidney or liver impairment.
* Moderate to severe asthma.
* Type I diabetes.
* Gastrointestinal illness.
* Use of any prescription or over-the-counter medication except birth control or non-steroidal antiinflammatory drugs on an as-needed basis.
* History of or current neurological illnesses, such as stroke, seizure disorders, neurodegenerative diseases, or organic brain syndrome.
* Learning disability, mental retardation, or any other condition that impedes cognition.
* Any surgeries requiring full anesthesia scheduled within 2 weeks of any of the study test sessions.
* Inability to perform the Rapid Visual Information Processing Task.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Spatial Attentional Resource Allocation Task reaction time | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  average reaction time of trials with a signal detection response
Spatial Attentional Resource Allocation Task omission errors | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  percentage of trials on which no response was registered
Rapid Visual Information Processing Task signal detection | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  signal detection index based on hit rate and false alarm rate
Rapid Visual Information Processing Task reaction time | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  average reaction time on trials with a correct response
Change Detection Task accuracy | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  % of correct responses
Change Detection reaction time | 5 hrs after patch application (=1 hr after ingestion of oral solution) on each test day
  average reaction time across trials

SECONDARY OUTCOMES:
Vital signs: blood pressure | hourly for 8 hours on each test day
  mm Hg
Vital signs: heart rate | hourly for 8 hours on each test day
  beats per minute
ECG | Before and 4 hours after ingestion of oral solution on each test day
  QTc interval

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available, in de-identified form, to Anvyl LLC (Irvine, CA).